CLINICAL TRIAL: NCT04209712
Title: Phase I Clinical Trial of Haploid Donor-derived in Vitro Activated Natural Killer Cells Infusion for Patients With Minimal Residual Disease After Consolidation Therapy for Acute Myeloid Leukemia
Brief Title: Natural Killer Cells Infusion for Treating Acute Myeloid Leukemia Patients With Minimal Residual Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Collaborators: Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS2019070101
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: haploid allogeneic NK cell therapy with chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- haploid allogeneic NK cell therapy (Experimental): haploid allogeneic NK cell therapy with chemotherapy
  Interventions: Biological: haploid allogeneic NK cell therapy

INTERVENTIONS:
Biological: haploid allogeneic NK cell therapy — NK cells will be intravenously infused to the patient for 2 days, with following subcutaneously injection of Interleukin-2.

SUMMARY:
This trial will evaluate the effectiveness and safety of haploid donor-derived in vitro activated natural killer(NK) cells infusion for Treating acute myeloid leukemia Patients With minimal residual disease.

DETAILED DESCRIPTION:
Patients of acute myeloid leukemia after chemotherapy with MRD(minimal residual disease) will receive NK cell infusion combined with consolidation chemotherapy. The bone marrow morphology and MRD remission of the patients will be observed 15 days after the same treatment. All patients will be followed up for 1 year.

NK cells are prepared in Beijing iCELL Biotechnology Co.,Ltd, which is subsidiary to Shanghai iCELL Biotechnology Co.,Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with acute myeloid leukemia;
2. MRD after 2 course of standard chemotherapy;
3. No plan for hematopoietic stem cell transplantation;
4. Hemoglobin (Hb) >=60g/L, white blood cell count (WBC) >=2.5x10^9/L, platelet count >=30x10^9/L;
5. Patients have self-knowledge ability and can sign informed and voluntary consent forms;
6. Patients or their clients, guardians of pediatric patients signed the informed and voluntary consent form and joined the study.

Exclusion Criteria:

1. Intracranial hypertension or unconsciousness;
2. Symptomatic heart failure or severe arrhythmia;
3. Respiratory failure;
4. With other types of malignant tumor diseases;
5. T lymphocytic acute leukemia;
6. Diffuse intravascular;
7. Serum creatinine and / or urea nitrogen >=1.5 times the normal value;coagulation;
8. Serum total bilirubin >=1.5 times the normal value;
9. Sepsis or other difficult-to-control infections;
10. Uncontrollable diabetes;
11. severe mental disorders;
12. WHO physical status classification >=3;
13. People who are allergic to Interleukin-2;
14. Patients after organ transplant;
15. Pregnant and lactating women.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease (MRD) | 12 months
  MRD-negative is defined as <0.1% blasts with leukemia-associated phenotype detected by flow cytometry. MRD-positive is defined as >=0.1% blasts with leukemia-associated phenotype detected by flow cytometry.

SECONDARY OUTCOMES:
Number of participants with adverse events | 12 months
  Evaluation of toxicities defined as any CTCAE (v. 4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Xian Zhang, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Langfang, Hebei, China